CLINICAL TRIAL: NCT03506399
Title: Effect of Lanabecestat on the Pharmacokinetics of Ethinyl Estradiol and Levonorgestrel in Healthy Female Subjects
Brief Title: A Study of Lanabecestat in Healthy Female Participants Taking Oral Contraceptive
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Stopped for futility. Phase 3 studies not likely to meet primary endpoints.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16004; I8D-MC-AZEK (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-04-20; First posted 2018-04-24 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Healthy
MeSH Terms: interventions — lanabecestat; Contraceptives, Oral; ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oral Contraceptive (OC) (Experimental): Ethinyl estradiol and levonorgestrel administered as a single dose, orally
  Interventions: Drug: Oral Contraceptive
- Lanabecestat (Experimental): Single oral dose of lanabecestat
  Interventions: Drug: Lanabecestat
- Lanabecestat and OC (Experimental): A single oral dose of oral contraceptive and single daily doses of lanabecestat
  Interventions: Drug: Lanabecestat; Drug: Oral Contraceptive

INTERVENTIONS:
Drug: Lanabecestat — Administered orally
  Other Names: LY3314814
  Arms: Lanabecestat; Lanabecestat and OC
Drug: Oral Contraceptive — Administered orally
  Other Names: Ethinyl Estradiol and Levonorgestrel
  Arms: Lanabecestat and OC; Oral Contraceptive (OC)

SUMMARY:
The study will evaluate the effect of oral contraceptive (birth control pill) on the blood level of lanabecestat when both are given together. Side effects will be monitored and documented. This study will last up to 27 days for each participant, not including screening. Screening is required within 42 days prior to first dose.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy female participants
* Women not of childbearing potential; women of childbearing potential using a non-hormonal intrauterine device (IUD)
* Have a body mass index (BMI) of 17.5 to 32 kilogram per meter square (kg/m²)

Exclusion Criteria:

* Have a history of or current significant ophthalmic disease, which includes participants with clinically significant eye abnormalities, particularly any eye problem involving the retina, as determined by the investigator
* Have vitiligo or any other clinically significant disorder of skin or hair pigmentation, as determined by the investigator
* Have a history of or current neuropsychiatric disease/condition including psychosis, affective disorder, anxiety disorder, borderline state, or personality disorder

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under The Concentration Curve (AUC) of Ethinyl Estradiol | Baseline though 120 hours after administration of the study drug (lanabecestat)
  PK: AUC of Ethinyl Estradiol
PK: AUC of Levonorgestrel | Baseline though 120 hours after administration of the study drug (lanabecestat)
  PK: AUC of Levonorgestrel
PK: Maximum Observed Concentration (Cmax) of Ethinyl Estradiol | Baseline though 120 hours after administration of the study drug (lanabecestat)
  PK: Cmax of Ethinyl Estradiol
PK: Cmax of Levonorgestrel | Baseline though 120 hours after administration of the study drug (lanabecestat)
  PK: Cmax of Levonorgestrel

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore